CLINICAL TRIAL: NCT05236738
Title: An Open-Label, Randomized, Single-Dose, 3-Treatment, 3-Period, 3-Sequence, Crossover Design, Relative Bioavailability Study Comparing the Pharmacokinetics of Atazanavir and Cobicistat Between the Coadministration of Age-Appropriate Mini-Tablet Formulations (ATV and COBI Oral Mini-tablets; 300 mg and 150 mg, Respectively) and the Coadministration of the Individual Reference Products (REYATAZ [Atazanavir Oral Powder] and TYBOST [Cobicistat Oral Tablet]; 300 mg and 150 mg, Respectively) in Healthy Adults Under Fed Conditions
Brief Title: A Study to Compare the Drug Levels of Atazanavir and Cobicistat Between the Coadministration of Age-Appropriate Mini-Tablet Formulations and the Coadministration of the Individual Reference Products in Healthy Adults Under Fed Conditions
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Bristol-Myers Squibb (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: AI424-578
Expanded Access: NCT00046345 (No longer available)
Record Dates: First submitted 2022-02-02; First posted 2022-02-11 (Actual); Last update posted 2022-10-31 (Actual); Status verified 2022-10

CONDITIONS: Healthy Participants
Keywords: Healthy Participants; Atazanavir; Cobicistat; Reyataz; Tybost; Evotaz
MeSH Terms: interventions — Atazanavir Sulfate; Cobicistat

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Treatment Sequence Group 1 (Experimental)
  Interventions: Drug: Atazanavir; Drug: Cobicistat; Drug: Atazanavir/Cobicistat Mini-tablet
- Treatment Sequence Group 2 (Experimental)
  Interventions: Drug: Atazanavir; Drug: Cobicistat; Drug: Atazanavir/Cobicistat Mini-tablet
- Treatment Sequence Group 3 (Experimental)
  Interventions: Drug: Atazanavir; Drug: Cobicistat; Drug: Atazanavir/Cobicistat Mini-tablet

INTERVENTIONS:
Drug: Atazanavir — Specified dose on specified days
  Other Names: ATV; Reyataz
Drug: Cobicistat — Specified dose on specified days
  Other Names: COBI; Tybost
Drug: Atazanavir/Cobicistat Mini-tablet — Specified dose on specified days
  Other Names: Evotaz

SUMMARY:
The purpose of this study is to evaluate the drug absorption of atazanavir and cobicistat between the coadministration of the mini-tablet formulations in applesauce or chocolate pudding followed by water and the coadministration of atazanavir oral powder in applesauce and cobicistat oral tablet followed by water in healthy adult participants.

ELIGIBILITY:
Inclusion Criteria:

• Body Mass Index (BMI) of 18.0 to 32.0 kg/m^2, inclusive. BMI = weight (kg)/[height(m)]^2

Exclusion Criteria:

* Significant acute or chronic medical illness
* History of a clinically significant drug rash, Stevens-Johnson Syndrome or Gilbert's Syndrome
* Inability to swallow oral medication
* Major surgery within 4 weeks of study treatment administration

Other protocol-defined inclusion/exclusion criteria apply

Ages: 18 Years to 49 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 42 (Actual)
Dates: Start 2022-05-13 (Actual); Primary Completion 2022-07-05 (Actual); Study Completion 2022-07-26 (Actual)

PRIMARY OUTCOMES:
Maximum observed plasma concentration (Cmax) | Up to 17 days
Area under the plasma concentration-time curve from time zero extrapolated to infinite time (AUC[INF]) | Up to 17 days

SECONDARY OUTCOMES:
Time of maximum observed plasma concentration (Tmax) | Up to 17 days
Apparent terminal plasma half-life (T-HALF) | Up to 17 days
Area under the plasma concentration-time curve from time zero to time of last quantifiable concentration (AUC[0-T]) | Up to 17 days
Observed plasma concentration at 24 hours (C24) | Up to 17 days
Number of participants with Adverse Events (AEs) | Up to 75 days
Number of participants with Serious Adverse Events (SAEs) | Up to 75 days
Number of participants with AEs leading to discontinuation | Up to 75 days
Number of participants with AEs leading to death | Up to 75 days
Number of participants with clinical laboratory abnormalities | Up to 17 days
Number of participants with vital sign abnormalities | Up to 17 days
Number of participants with electrocardiogram (ECG) abnormalities | Up to 17 days
Changes in Taste Evaluation Questionnaire | Up to 17 days
  Palatability evaluated on a scale from 1 (weak) to 9 (strong)

CONTACTS AND LOCATIONS:
Overall Officials: Bristol-Myers Squibb, Study Director — Bristol-Myers Squibb
Locations (1):
- Local Institution - 0001, Miami, Florida, United States

REFERENCES:
- See also: BMS Clinical Trial Information — https://www.bms.com/researchers-and-partners/clinical-trials-and-research.html
- See also: BMS Clinical Trial Patient Recruiting — https://www.bmsstudyconnect.com/s/US/English/USenHome
- See also: Investigator Inquiry Form — https://www.bms.com/researchers-and-partners/clinical-trials-and-research.html
- See also: FDA Safety Alerts and Recalls — https://www.fda.gov/Safety/MedWatch/SafetyInformation/default.htm